CLINICAL TRIAL: NCT01566539
Title: The Biological Basis of Individual Variation in Social Cooperation
Brief Title: Biological Basis of Individual Variation in Social Cooperation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); John Templeton Foundation (Other)
Responsible Party: Principal Investigator, James K. Rilling, PhD, Associate Professor, Emory University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00007905; 1R01MH084068-01A1 (NIH); MH087721-01A1 (Other: NIMH)
Record Dates: First submitted 2012-03-26; First posted 2012-03-29 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: Social cooperation; Oxytocin; Vasopressin; Prisoner's Dilemma game; Empathy; fMRI
MeSH Terms: conditions — Diabetes Insipidus | interventions — Lorazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (11):
- Healthy Volunteers - Intranasal Vasopressin (AVP) (Experimental): The AVP group of healthy volunteers will self-administer vasopressin solution prior to completing the PD task.
  Interventions: Drug: Intranasal Vasopressin (AVP)
- Healthy Volunteers - Intranasal Oxytocin (OT) (Experimental): The OT group of healthy volunteers will self-administer oxytocin solution prior to completing the PD task.
  Interventions: Drug: Intranasal Oxytocin (OT) 24 IU
- Healthy Volunteers - Intranasal Placebo (Placebo Comparator): The placebo group of healthy volunteers will self-administer a placebo spray prior to completing the PD task.
  Interventions: Drug: Intranasal Placebo
- Within Subject Group (Experimental): Some healthy volunteer participants who received drug in their first session will receive placebo in their second session and vice-versa prior to completing the PD task. For each gender, half will receive AVP in one session and placebo in the other session, and half will receive OT in one session and placebo in the second session. In each group, half of the subjects will receive drug first and half will receive placebo first. Additionally, a group of subjects who receive placebo the first time will receive placebo the second time.
  Interventions: Drug: Intranasal Oxytocin (OT) 24 IU; Drug: Intranasal Vasopressin (AVP); Drug: Intranasal Placebo
- Faces Task - Vasopressin (AVP) (Experimental): Healthy volunteers between the ages of 21-30 years will receive Faces Intranasal Vasopressin (AVP) prior to completing the Faces task during fMRI scanning.
  Interventions: Drug: Intranasal Vasopressin (AVP) 40 IU
- Faces Task - Placebo (Placebo Comparator): Healthy volunteers between the ages of 21-30 years will receive placebo prior to completing the Faces task during fMRI scanning.
  Interventions: Drug: Intranasal Placebo
- Empathy Task - Oxytocin (OT) (Experimental): Healthy volunteers between the ages of 18-30 years will receive placebo at scan 1 and OT at scan 2 prior to completing an empathy task.
  Interventions: Drug: Intranasal Oxytocin (OT) 24 IU; Drug: Intranasal Placebo
- Empathy Task - Placebo (Placebo Comparator): Healthy volunteers between the ages of 18-30 years will receive placebo at scan 1 and placebo at scan 2 prior to completing an empathy task.
  Interventions: Drug: Intranasal Placebo
- Anxious and Depressed Subjects - OT (Experimental): Depressed or anxious men between the ages of 18 and 22 will receive intranasal OT prior to completing the Prisoner's Dilemma game task and MRI scan.
  Interventions: Drug: Intranasal Oxytocin (OT) 24 IU
- Anxious and Depressed Subjects - Placebo (Placebo Comparator): Depressed or anxious men between the ages of 18 and 22 will receive intranasal placebo prior to completing the Prisoner's Dilemma game task and MRI scan.
  Interventions: Drug: Intranasal Placebo
- Healthy Volunteers - Lorazepam (Experimental): Healthy normal men between the ages of 18 and 22 will receive lorazepam prior to completing the Prisoner's Dilemma game task and MRI scan.
  Interventions: Drug: Lorazepam

INTERVENTIONS:
Drug: Intranasal Oxytocin (OT) 24 IU — Participants will self-administer a single dose of 24 international units (IU) oxytocin. Five puffs per nostril, each with 2.4 IU oxytocin. Ten puffs total.
  Other Names: Oxytocin: Syntocinon Nasal Spray
  Arms: Anxious and Depressed Subjects - OT; Empathy Task - Oxytocin (OT); Healthy Volunteers - Intranasal Oxytocin (OT); Within Subject Group
Drug: Intranasal Vasopressin (AVP) — Participants will self-administer a 1 ml solution containing 20 units of AVP. Five puffs per nostril, each with 2 International Units (IU) AVP. Ten puffs total).
  Arms: Healthy Volunteers - Intranasal Vasopressin (AVP); Within Subject Group
Drug: Intranasal Placebo — Participants will receive placebo sprays that are pH adjusted to comparable levels of the drugs given. Five puffs per nostril; ten puffs total.
  Arms: Anxious and Depressed Subjects - Placebo; Empathy Task - Oxytocin (OT); Empathy Task - Placebo; Faces Task - Placebo; Healthy Volunteers - Intranasal Placebo; Within Subject Group
Drug: Intranasal Vasopressin (AVP) 40 IU — Participants will self-administer a 0.5 ml solution containing 40 international units (IU) of AVP. 5 puffs in total, each with 4 International Units (IU) AVP.
  Arms: Faces Task - Vasopressin (AVP)
Drug: Lorazepam — Subjects will take 1.0 mg of lorazepam orally 60 minutes prior to fMRI scan.
  Arms: Healthy Volunteers - Lorazepam

SUMMARY:
The project has three overall objectives. The first is to determine whether and how administration of intranasal oxytocin (OT) and intranasal vasopressin (AVP) influence cooperative decision-making and neural responses to cooperative and un-cooperative social interactions. The second is to determine whether and how intranasal vasopressin influences subjective evaluations of and neural responses to same and opposite-sex face stimuli and to determine if any of these effects persist beyond the period of AVP exposure. The third objective is to determine if intranasal OT influences empathy-related behavior and associated brain activity.

DETAILED DESCRIPTION:
There are several objective to the study.

Objective 1: In this double-blind, placebo-controlled, pharmaco- fMRI study, men and women will be randomized to treatment with either 24 IU intranasal OT, 20 IU intranasal AVP, or placebo (PL). Approximately 40 minutes later, brain function will be imaged with fMRI as participants play an iterated Prisoner's Dilemma game with same-sex partners. The resulting data will be analyzed to investigate OT and AVP effects on cooperative behavior and the neural response to cooperative social interactions.

In addition to this cross-sectional design, a subset of participants will return on a second day for a within-subject study.

Objective 2: Men and healthy women will be randomized to treatment with either 40 IU intranasal AVP or a saline placebo approximately 30 minutes before their brain function is measured with fMRI as they view same and other-sex faces. All subjects will be scanned a second time several days later with no treatment to evaluate the persistence of AVP effects over time. The resulting data will be analyzed to investigate AVP effects on subjective evaluations and neural responses to viewing same and opposite sex faces.

Objective 3: Healthy men and healthy women will receive either 24IU intranasal OT or PL approximately 40 minutes before their brain function is measured with fMRI as they view animations of geometric shapes depicting either random movement or social interactions such as playing, chasing, fighting. All participants will receive PL on scan 1 and will be randomized to either 24IU intranasal OT or PL on scan 2. The resulting data will be analyzed to investigate OT effects on subjective evaluations and neural responses to the animations.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years of age
* 21-30 for Faces component
* Normal or corrected-to-normal vision of 20/40
* Unmedicated depressed or anxious men between 18-22 years of age for Anxious and Depressed component

Exclusion Criteria:

* Pregnancy, recent birth, or breastfeeding
* History of seizures
* Neurological Disorder
* Current psychiatric disorder
* Previous psychiatric disorder (can be included as discretion of PI)
* Current use of psychoactive drugs
* Previous use of psychoactive drugs (can be included as discretion of PI)
* Previous head trauma (can be included at discretion of PI)
* Alcoholism or substance abuse
* Hypertension
* Cardiovascular Disease
* Nephritis
* Diabetes
* Endocrine disease or malignancy
* Asthma (can be included as discretion of PI, if episodes are infrequent, nonmedicated, and no active problems at time of study)
* Migraines (can be included as discretion of PI, if episodes are infrequent, nonmedicated, and no active problems at time of study)
* Claustrophobia (at discretion of PI)

Additional exclusion criteria for Lorazepam arm

* Acute narrow-angle glaucoma
* Compromised respiratory function (e.g. sleep apnea and chronic obstructive pulmonary disease)
* Impaired renal and hepatic function

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 707 (Actual)
Dates: Start 2008-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James K Rilling, Ph.D., Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital, Atlanta, Georgia
  - Emory University 1462 Clifton Rd, Atlanta, Georgia

REFERENCES:
- [Background] Kosfeld M, Heinrichs M, Zak PJ, Fischbacher U, Fehr E. Oxytocin increases trust in humans. Nature. 2005 Jun 2;435(7042):673-6. doi: 10.1038/nature03701. PMID 15931222
- [Background] Fisher H, Aron A, Brown LL. Romantic love: an fMRI study of a neural mechanism for mate choice. J Comp Neurol. 2005 Dec 5;493(1):58-62. doi: 10.1002/cne.20772. PMID 16255001
- [Background] Thompson RR, George K, Walton JC, Orr SP, Benson J. Sex-specific influences of vasopressin on human social communication. Proc Natl Acad Sci U S A. 2006 May 16;103(20):7889-94. doi: 10.1073/pnas.0600406103. Epub 2006 May 8. PMID 16682649
- [Background] Vrticka P, Andersson F, Sander D, Vuilleumier P. Memory for friends or foes: the social context of past encounters with faces modulates their subsequent neural traces in the brain. Soc Neurosci. 2009;4(5):384-401. doi: 10.1080/17470910902941793. Epub 2009 Jul 27. PMID 19637101
- [Background] Singer T, Kiebel SJ, Winston JS, Dolan RJ, Frith CD. Brain responses to the acquired moral status of faces. Neuron. 2004 Feb 19;41(4):653-62. doi: 10.1016/s0896-6273(04)00014-5. PMID 14980212
- [Background] Guroglu B, Haselager GJ, van Lieshout CF, Takashima A, Rijpkema M, Fernandez G. Why are friends special? Implementing a social interaction simulation task to probe the neural correlates of friendship. Neuroimage. 2008 Jan 15;39(2):903-10. doi: 10.1016/j.neuroimage.2007.09.007. Epub 2007 Sep 15. PMID 17964185
- See also: Related Info — http://anthropology.emory.edu/home/people/faculty/rilling.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 707 signed the consent form, 449 started the main study period.
Pre-assignment Details: The study team did not recruit any participants for the "Anxious and Depressed Subjects - OT", or "Anxious and Depressed Subjects - Placebo" arms.Therefore, these arms have been removed from the record.
Groups:
- Within Subject Group: Some healthy volunteer participants who received drug in their first session will receive placebo in their second session and vice-versa prior to completing the PD task. For each gender, half will receive AVP in one session and placebo in the other session, and half will receive OT in one session and placebo in the second session. In each group, half of the subjects will receive drug first and half will receive placebo first. Additionally, a group of subjects who receive placebo the first time will receive placebo the second time.
  Intranasal Oxytocin (OT) 24 IU: Participants will self-administer a single dose of 24 international units (IU) oxytocin. Five puffs per nostril, each with 2.4 IU oxytocin. Ten puffs total.
  Intranasal Vasopressin (AVP): Participants will self-administer a 1 ml solution containing 20 units of AVP. Five puffs per nostril, each with 2 International Units (IU) AVP. Ten puffs total).
  Intranasal Placebo: Participants will receive placebo sprays that are pH
Period: Main Study Period
Arm/Group | Healthy Volunteers - Intranasal Vasopressin (AVP) | Healthy Volunteers - Intranasal Oxytocin (OT) | Healthy Volunteers - Intranasal Placebo | Within Subject Group | Faces Task - Vasopressin (AVP) | Faces Task - Placebo | Empathy Task - Oxytocin (OT) | Empathy Task - Placebo | Healthy Volunteers - Lorazepam
Started | 101 | 100 | 104 | 0 | 40 | 43 | 30 | 30 | 1
Completed | 100 | 100 | 104 | 0 | 40 | 40 | 30 | 30 | 1
Not Completed | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Period: Within Subject Group
Arm/Group | Healthy Volunteers - Intranasal Vasopressin (AVP) | Healthy Volunteers - Intranasal Oxytocin (OT) | Healthy Volunteers - Intranasal Placebo | Within Subject Group | Faces Task - Vasopressin (AVP) | Faces Task - Placebo | Empathy Task - Oxytocin (OT) | Empathy Task - Placebo | Healthy Volunteers - Lorazepam
Started | 0 | 0 | 0 | 156 (Participants can move from Healthy Volunteers-AVP, OT and Placebo groups to the within subject group) | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 153 (Participants can move from Healthy Volunteers-AVP, OT and Placebo groups to the within subject group) | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers - Intranasal Vasopressin (AVP) | Healthy Volunteers - Intranasal Oxytocin (OT) | Healthy Volunteers - Intranasal Placebo | Faces Task - Vasopressin (AVP) | Faces Task - Placebo | Empathy Task - Oxytocin (OT) | Empathy Task - Placebo | Healthy Volunteers - Lorazepam | Total
Number analyzed (Participants) | 101 | 100 | 104 | 40 | 43 | 30 | 30 | 1 | 449
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 101 | 100 | 104 | 40 | 43 | 30 | 30 | 1 | 449
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 50 | 50 | 20 | 21 | 15 | 15 | 0 | 223
  Male | 49 | 50 | 54 | 20 | 22 | 15 | 15 | 1 | 226
Region of Enrollment [Number; unit: participants]
  United States | 101 | 100 | 104 | 40 | 43 | 30 | 30 | 1 | 449

OUTCOME MEASURES:

1. Primary Outcome: Healthy Volunteers-OT, Placebo: Mean Percent Signal Change in Right Caudate Nucleus in Men
Description: The effect of the drug treatment will be assessed by determining differences in brain activation between OT and placebo groups in the right caudate nucleus region during reciprocated cooperation in Prisoner Dilemma game while undergoing an fMRI scan.
Time Frame: Visit 1 (40-100 Minutes Post-Intervention)
Population: Analysis was completed in the Healthy Volunteers - Intranasal Oxytocin (OT) and Healthy Volunteers - Intranasal Placebo groups per protocol. Subjects with excessive motion, missing data, abnormal brain anatomy or partial data collection were excluded from the analysis.
Measure: Mean (Standard Error); unit: percent signal change
Arm/Group | Healthy Volunteers - Intranasal Oxytocin (OT) | Healthy Volunteers - Intranasal Placebo
Number analyzed (Participants) | 43 | 48
percent signal change | 0.21 (0.03) | 0.07 (0.02)

2. Primary Outcome: Healthy Volunteers-OT, Placebo: Mean Percent Signal Change in Right Caudate Nucleus in Women
Description: as for outcome 1
Time Frame: Visit 1 (40-100 Minutes Post-Intervention)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percent signal change
Arm/Group | Healthy Volunteers - Intranasal Oxytocin (OT) | Healthy Volunteers - Intranasal Placebo
Number analyzed (Participants) | 47 | 46
percent signal change | 0.04 (0.02) | 0.15 (0.02)

3. Primary Outcome: Healthy Volunteers-AVP, Placebo: Mean Percent Signal Change in Left Insula in Men
Description: The effect of the drug treatment will be assessed by determining differences in brain activation between AVP and placebo groups in the left insula region during reciprocated cooperation in Prisoner Dilemma game while undergoing an fMRI scan.
Time Frame: Visit 1 (40-100 Minutes Post-Intervention)
Population: Analysis was completed in the Healthy Volunteers - Intranasal Vasopressin (AVP) and Healthy Volunteers - Intranasal Placebo groups per protocol. Subjects with excessive motion, missing data, abnormal brain anatomy or partial data collection were excluded from the analysis.
Measure: Mean (Standard Error); unit: percent signal change
Arm/Group | Healthy Volunteers - Intranasal Vasopressin (AVP) | Healthy Volunteers - Intranasal Placebo
Number analyzed (Participants) | 44 | 48
percent signal change | 0.13 (0.02) | -0.02 (0.02)

4. Primary Outcome: Healthy Volunteers-AVP, Placebo: Mean Percent Signal Change in Left Insula in Women
Description: The effect of the drug treatment will be assessed by determining differences in brain activation between AVP and placebo groups in the left insula during reciprocated cooperation in Prisoner Dilemma game while undergoing an fMRI scan.
Time Frame: Visit 1 (40-100 Minutes Post-Intervention)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: percent signal change
Arm/Group | Healthy Volunteers - Intranasal Vasopressin (AVP) | Healthy Volunteers - Intranasal Placebo
Number analyzed (Participants) | 49 | 46
percent signal change | -0.05 (0.03) | 0.10 (0.03)

5. Primary Outcome: Within Subject Group: Mean Percent Signal Change in Left Caudate Nucleus in Men and Women
Description: The effect of the drug will be assessed by determining changes in brain activation between the visit where the participant received drug and the visit where the participant received PL in the right caudate during reciprocated cooperation in Prisoner Dilemma game while undergoing an fMRI scan.
Time Frame: Visit 1 (30-75 Minutes Post-Intervention), Visit 2 (Up to 2 Weeks)
Population: Analysis was completed for the within subject group per protocol. Subjects with excessive motion during scanning were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percent signal change
Arm/Group | Within Subject Group
Number analyzed (Participants) | 57
percent signal change
  Oxytocin treatment in men | 0.21 (0.19)
  Placebo treatment in men | 0.19 (0.29)
  Oxytocin treatment in women | 0.06 (0.21)
  Placebo treatment in women | 0.10 (0.18)

6. Secondary Outcome: Healthy Volunteer Groups: Total Number of Cooperate Choices Made by Men During the Prisoners Dilemma Game
Description: The effect of the drug treatments will be assessed by determining the number of cooperative choices made during the prisoner's dilemma game. Participants may make two choices that are considered "cooperative". The higher the total number, the more cooperative choices made.
Time Frame: Visit 1 (40-100 Minutes Post-Intervention)
Population: Analysis was completed for the Healthy Volunteers - Intranasal Vasopressin (AVP), Healthy Volunteers - Intranasal Oxytocin (OT), and Healthy Volunteers - Intranasal Placebo groups per protocol. Subjects with missing data were excluded from the analysis.
Measure: Mean (Standard Error); unit: number of choices
Arm/Group | Healthy Volunteers - Intranasal Vasopressin (AVP) | Healthy Volunteers - Intranasal Oxytocin (OT) | Healthy Volunteers - Intranasal Placebo
Number analyzed (Participants) | 49 | 50 | 53
number of choices | 15.71 (0.98) | 16.18 (1.01) | 17.68 (0.93)

7. Secondary Outcome: Healthy Volunteer Groups: Total Number of Cooperate Choices Made by Women During the Prisoners Dilemma Game
Description: as for outcome 6
Time Frame: Visit 1 (40-100 Minutes Post-Intervention)
Population: as for outcome 6
Measure: Mean (Standard Error); unit: number of choices
Arm/Group | Healthy Volunteers - Intranasal Vasopressin (AVP) | Healthy Volunteers - Intranasal Oxytocin (OT) | Healthy Volunteers - Intranasal Placebo
Number analyzed (Participants) | 51 | 50 | 50
number of choices | 15.84 (0.76) | 18.14 (1.03) | 16.92 (0.98)

8. Secondary Outcome: Within Subject Group: Mean Difference in Number of Cooperate Choices Made by Male During the Prisoners Dilemma Game
Description: as for outcome 6
Time Frame: Visit 1 (30-75 Minutes Post-Intervention), Visit 2 (Up to 2 Weeks)
Population: Analysis was completed for the Within Subject Group per protocol. Subjects with missing data were excluded from the analysis. The difference between OT and PL visits is reported here (OT-PL).
Measure: Mean (Standard Deviation); unit: number of choices
Arm/Group | Within Subject Group
Number analyzed (Participants) | 29
number of choices | -1.10 (5.21)

9. Secondary Outcome: Within Subject Group: Mean Difference in Number of Cooperate Choices Made by Female During the Prisoners Dilemma Game
Description: as for outcome 6
Time Frame: Visit 1 (30-75 Minutes Post-Intervention), Visit 2 (Up to 2 Weeks)
Population: Analysis was completed for the Within Subject Group per protocol. Subjects with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: number of choices
Arm/Group | Within Subject Group
Number analyzed (Participants) | 30
number of choices
  Oxytocin treatment | 16.13 (6.87)
  Placebo treatment | 15.53 (6.70)

10. Secondary Outcome: Faces Task Groups: Mean Percent Signal Change in Nucleus Accumbens to Faces in Men
Description: The effect of the drug treatment will be assessed by determining differences in brain activation between AVP and PL group when participants are viewing same-sex faces, and when participants are viewing other-sex faces.
Time Frame: Visit 1 (30-75 Minutes Post-Intervention), Visit 2 (Up to 7 Days)
Population: Analysis was completed for the Faces Task - Vasopressin (AVP) and Faces Task - Placebo groups per protocol. Subjects with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percent signal change
Arm/Group | Faces Task - Vasopressin (AVP) | Faces Task - Placebo
Number analyzed (Participants) | 20 | 20
percent signal change
  viewing same-sex faces | 0.03 (0.30) | -0.14 (0.22)
  viewing other-sex faces | 0.14 (0.33) | -0.13 (0.30)

11. Secondary Outcome: Faces Task Groups: Mean Percent Signal Change in Nucleus Accumbens to Faces in Women
Description: as for outcome 10
Time Frame: Visit 1 (30-75 Minutes Post-Intervention), Visit 2 (Up to 7 Days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percent signal change
Arm/Group | Faces Task - Vasopressin (AVP) | Faces Task - Placebo
Number analyzed (Participants) | 20 | 19
percent signal change
  viewing same-sex faces | -0.08 (0.31) | 0.12 (0.22)
  viewing other-sex faces | 0.003 (0.16) | 0.13 (0.22)

12. Secondary Outcome: Faces Task Groups: Mean Approachability Rating of Faces in Men
Description: Approachability is rated by a study specific seven point scale where -3 indicates threatening and unapproachable and +3 indicates friendly and approachable. Participants will rate same-sex and other-sex faces. The effect of the drug treatment will be assessed by determining differences in approachability ratings between AVP and PL group when participants are viewing same-sex faces, and when participants are viewing other-sex faces.
Time Frame: Visit 1 (30-75 Minutes Post-Intervention), Visit 2 (Up to 7 Days)
Population: Data was collected per protocol in the AVP and placebo faces groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Faces Task - Vasopressin (AVP) | Faces Task - Placebo
Number analyzed (Participants) | 20 | 20
units on a scale
  viewing same-sex faces scan 1 | 0.31 (0.96) | -0.06 (0.96)
  viewing other-sex faces scan 1 | 1.00 (1.09) | 0.81 (0.92)
  viewing same-sex faces scan 2 | 0.78 (0.88) | 0.25 (0.99)
  viewing other-sex faces scan 2 | 1.19 (1.04) | 0.89 (0.98)

13. Secondary Outcome: Faces Task Group: Mean Approachability Rating of Faces in Women
Description: as for outcome 12
Time Frame: Visit 1 (30-75 Minutes Post-Intervention), Visit 2 (Up to 7 Days)
Population: Data was collected per protocol in the AVP and placebo faces groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Faces Task - Vasopressin (AVP) | Faces Task - Placebo
Number analyzed (Participants) | 20 | 20
units on a scale
  viewing same-sex faces scan 1 | 0.37 (0.57) | 0.21 (0.86)
  viewing other-sex faces scan 1 | -0.04 (0.83) | 0.28 (0.61)
  viewing same-sex faces scan 2 | 0.37 (0.57) | 0.23 (0.88)
  viewing other-sex faces scan 2 | 0.12 (0.66) | 0.22 (0.63)

14. Secondary Outcome: Faces Task Groups: Mean Attractiveness Rating of Faces in Men
Description: Attractiveness is rated by a study specific seven point scale where -3 indicates least attractive and +3 indicates most attractive. Participants will rate same-sex and other-sex faces. The effect of the drug treatment will be assessed by determining differences in attractiveness ratings between AVP and PL group when participants are viewing same-sex faces, and when participants are viewing other-sex faces.
Time Frame: Visit 1 (30-75 Minutes Post-Intervention), Visit 2 (Up to 7 Days)
Population: Data was collected per protocol in the AVP and placebo faces groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Faces Task - Vasopressin (AVP) | Faces Task - Placebo
Number analyzed (Participants) | 20 | 20
units on a scale
  viewing same-sex faces scan 1 | 0.35 (0.78) | -0.06 (0.77)
  viewing other-sex faces scan 1 | 1.79 (0.58) | 1.60 (0.46)
  viewing same-sex faces scan 2 | 0.52 (0.86) | -0.08 (0.79)
  viewing other-sex faces scan 2 | 1.70 (0.69) | 1.43 (0.64)

15. Secondary Outcome: Faces Task Groups: Mean Attractiveness Rating of Faces in Women
Description: as for outcome 14
Time Frame: Visit 1 (30-75 Minutes Post-Intervention), Visit 2 (Up to 7 Days)
Population: Data was collected per protocol in the AVP and placebo faces groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Faces Task - Vasopressin (AVP) | Faces Task - Placebo
Number analyzed (Participants) | 20 | 20
units on a scale
  viewing same-sex faces scan 1 | 1.56 (0.54) | 1.02 (0.80)
  viewing other-sex faces scan 1 | 0.55 (1.16) | 0.61 (0.62)
  viewing same-sex faces scan 2 | 1.29 (0.68) | 0.82 (0.92)
  viewing other-sex faces scan 2 | 0.53 (1.04) | 0.28 (0.51)

16. Secondary Outcome: Empathy Task Groups: Mean Percent Signal Change in Early Visual Cortex in Response to Animation in Women
Description: The effect of the drug treatment will be assessed by determining differences in brain activation between OT and PL group when participants are viewing animations.
Time Frame: Visit 1 (40-75 Minutes Post-Intervention), Visit 2 (Up to 1 Month)
Population: Data was collected per protocol in the OT and placebo empathy task groups.
Measure: Mean (Standard Deviation); unit: percent signal change
Arm/Group | Empathy Task - Oxytocin (OT) | Empathy Task - Placebo
Number analyzed (Participants) | 15 | 15
percent signal change | -.910 (.417) | -.377 (.656)

17. Secondary Outcome: Empathy Task Groups: Mean Percent Signal Change in Early Visual Cortex in Response to Animation in Men
Description: as for outcome 16
Time Frame: Visit 1 (40-75 Minutes Post-Intervention), Visit 2 (Up to 1 Month)
Population: Data was collected per protocol in the OT and placebo empathy task groups.
Measure: Mean (Standard Deviation); unit: percent signal change
Arm/Group | Empathy Task - Oxytocin (OT) | Empathy Task - Placebo
Number analyzed (Participants) | 15 | 15
percent signal change | -.429 (.711) | -.382 (1.012)

18. Other Pre Specified Outcome: Healthy Volunteers Groups: Mean Vasopressin (AVP) Plasma Level
Description: Peripheral levels of AVP will be assessed via assay of plasma collected.
Time Frame: Visit 1 (Up to 3 Hours)
Population: Analysis was completed in the Healthy Volunteers - Intranasal Vasopressin (AVP), Healthy Volunteers - Intranasal Oxytocin (OT), and Healthy Volunteers - Intranasal Placebo groups per protocol. Subjects with unreliable or missing data were excluded from the analysis.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Healthy Volunteers - Intranasal Vasopressin (AVP) | Healthy Volunteers - Intranasal Oxytocin (OT) | Healthy Volunteers - Intranasal Placebo
Number analyzed (Participants) | 27 | 27 | 36
pg/ml | 4.5 (0.49) | 3.5 (0.34) | 3.1 (0.40)

19. Other Pre Specified Outcome: Healthy Volunteers Groups: Mean Oxytocin (OT) Plasma Level
Description: Peripheral levels of OT will be assessed via assay of plasma collected.
Time Frame: Visit 1 (Up to 3 Hours)
Population: as for outcome 18
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Healthy Volunteers - Intranasal Vasopressin (AVP) | Healthy Volunteers - Intranasal Oxytocin (OT) | Healthy Volunteers - Intranasal Placebo
Number analyzed (Participants) | 27 | 27 | 36
pg/ml | 120.6 (7.3) | 134.7 (10.2) | 129.4 (12.2)

20. Other Pre Specified Outcome: Healthy Volunteers Groups: Mean Testosterone Plasma Level
Description: Peripherals levels of testosterone will be assessed via assay of plasma collected.
Time Frame: Visit 1 (Up to 3 Hours)
Population: Analysis was completed in the first batch of data collection from Healthy Volunteers - Intranasal Vasopressin (AVP), Healthy Volunteers - Intranasal Oxytocin (OT), and Healthy Volunteers - Intranasal Placebo groups per protocol. Due to the lack of funds, no subsequent analysis has been done on the samples collected.
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Healthy Volunteers - Intranasal Vasopressin (AVP) | Healthy Volunteers - Intranasal Oxytocin (OT) | Healthy Volunteers - Intranasal Placebo
Number analyzed (Participants) | 25 | 30 | 31
ng/dl | 214.92 (125.42) | 475.82 (134.76) | 437.99 (160.36)

ADVERSE EVENTS:
Time Frame: Adverse event were collected throughout the duration of the study.
Arm/Group | Healthy Volunteers - Intranasal Vasopressin (AVP) | Healthy Volunteers - Intranasal Oxytocin (OT) | Healthy Volunteers - Intranasal Placebo | Within Subject Group | Faces Task - Vasopressin (AVP) | Faces Task - Placebo | Empathy Task - Oxytocin (OT) | Empathy Task - Placebo | Healthy Volunteers - Lorazepam
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/100 | 0/104 | 0/156 | 0/40 | 0/43 | 0/30 | 0/30 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/100 | 0/104 | 0/156 | 0/40 | 0/43 | 0/30 | 0/30 | 0/1
Other Adverse Events (participants affected / at risk) | 3/101 | 4/100 | 12/104 | 0/156 | 0/40 | 1/43 | 0/30 | 0/30 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteers - Intranasal Vasopressin (AVP) (N=101) | Healthy Volunteers - Intranasal Oxytocin (OT) (N=100) | Healthy Volunteers - Intranasal Placebo (N=104) | Within Subject Group (N=156) | Faces Task - Vasopressin (AVP) (N=40) | Faces Task - Placebo (N=43) | Empathy Task - Oxytocin (OT) (N=30) | Empathy Task - Placebo (N=30) | Healthy Volunteers - Lorazepam (N=1)
claustrophobia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — participants have claustrophobia and cannot enter a MRI scanner
fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Participant came in with a fever and was scheduled for later date. No procedures were done to the participant.
high blood pressure or heart rate post-drug administration (Vascular disorders) | 3 (3) | 3 (3) | 9 (9) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Subjects experience high blood pressure (above 140/90) or heart rate (above 100 bpm) post drug administration. Per protocol, subjects rested for 5-10 minutes and blood pressure and heart rate was retaken. They returned normal. Study proceeded.
felt faint after blood draw (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — subject felt faint after first blood draw. After resting, subject recovered and the study continued.
nose bleed (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — subject experience nose bleed prior to drug administration, probably due to dry weather.
nausea (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Subject experience nausea after drug administration.The subject believed it was due to hunger. Study physician was contacted and subject was provided some food. Once fed, the nausea subsided. He reported no side-effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes